CLINICAL TRIAL: NCT04985448
Title: Real World Study of the Effectiveness and Safety of Conbercept Ophthalmic Injection in the Treatment of Retinopathy of Prematurity - Multicenter, Retrospective and Observational Study Based on Real World Data
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Chengdu Kanghong Biotech Co., Ltd. (Industry)
Collaborators: Guangzhou Keli Medical Research Co., Ltd. (Unknown)
Responsible Party: Sponsor
Other Study IDs: KH902-ROP-CRP-2.0
Record Dates: First submitted 2021-07-23; First posted 2021-08-02 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Retinopathy of Prematurity
MeSH Terms: conditions — Retinopathy of Prematurity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Conbercept: In clinical treatment and research, the applied doses of Conbercept in patients with retinopathy of prematurity have been reduced compared with adults, mostly half of the adult dose. The commonly used exposure dose of intravitreal injection of Conbercept ophthalmic injection is 0.25mg/0.025ml.In addition, possible exposure doses are but not limited to 0.15mg/0.15ml, 0.1mg/ 0.1ml, 0.2mg/0.2ml, etc.
- Ranibizumab: In clinical treatment and research, the applied doses of Ranibizumab in patients with retinopathy of prematurity have been reduced compared with adults, mostly half of the adult dose. The commonly used exposure dose of intravitreal injection of Ranibizumab ophthalmic injection is 0.25mg/0.025ml.In addition, possible exposure doses are but not limited to 0.15mg/0.15ml, 0.1mg/ 0.1ml, 0.2mg/0.2ml, etc.
- Laser Treatment: In clinical and research studies, lasers are used to treat patients with retinopathy of prematurity.

SUMMARY:
This study is a retrospective, multi-center real world study. The real world data comes from the electronic medical record system and disease database of the research centers .The patient's demographic information, disease information, clinical treatment status, efficacy evaluation and adverse events and so on will be collected and evaluated by applicability of the data, generated an analysis data set. Use the causal inference method of statistical analysis to observe the effectiveness and safety of intravitreal injection of Conbercept, and explore the effectiveness and safety of different doses in the treatment of retinopathy of prematurity.

ELIGIBILITY:
Inclusion criteria:

1. Patient who are diagnosed as retinopathy of prematurity using clinical fundus screening;
2. Patients at the initial stage of treatment whose one eye at least has the following condition: Stage 1+, Stage 2+, Stage 3, Stage 3+ in Zone 1; or Stage 2+, Stage 3+ in Zone 2; or those with AP-ROP according to the international ROP classification,;
3. Patient for whom the first treatment is laser therapy, intravitreal injection of Conbercept or ranibizumab;

Exclusion criteria:

1. Patients with neurological diseases that seriously affect visual function;
2. Patient or his mother (during pregnancy) has received intravitreal or systemic anti-VEGF drug therapy for other diseases;

Elimination criteria:

1. Patients with insufficient data on treatment or medication;
2. Patients who are followed up for less than 3 months after treatment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients with retinopathy of prematurity in treatment of zone 1 (stage 1+, stage 2+, stage 3, stage 3+) or zone 2 (stage 2+, stage 3+) or AP-ROP (rapidly progressive posterior retinopathy of prematurity)
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Main effectiveness indicators | 24 weeks
  Proportion of eyes with no active retinopathy of prematurity and no structural adverse outcome (within 24 weeks after the first treatment; active retinopathy of prematurity is defined as additional lesions, vascular tortuosity, crest and other lesions having no alleviation but trend of progress after clinical treatment and new blood vessels continuing to exist or new born; poor structural outcomes are defined as adverse results such as retinal detachment, retinal traction or macular abnormalities after clinical treatment)
Main safety indicators | 24weeks
  The proportion of affected eyes with ocular AEs (within 24 weeks after the first treatment)
Primary endpoint | 24 weeks
  To evaluate the proportion of eyes with inactive retinopathy of prematurity and without structural adverse outcomes at 24 weeks after the first treatment (inactive retinopathy of prematurity is defined as the reduction in additional lesions, vascular tortuosity, ridges and other lesions after clinical treatment, showing no trend of progression, no persistent or newly developed neovascularization; no structural adverse outcome is defined as the absence of adverse outcomes such as retinal detachment, retinal traction, or macular abnormalities after clinical treatment)

SECONDARY OUTCOMES:
Secondary endpoints | at 1 week and 24 weeks
  To evaluate the response rate of the first treatment at 1 week and 24 weeks after the first treatment (the response rate is defined as the proportion of patients after the first treatment who do not need the second treatment, with disappearance of the additional lesions or the reduction of the vascular tortuosity, the reduction or regression of the ridges, and with initiation of vascularization in the neighboring avas-cular area (or retinal vascularization to zone III);
Secondary endpoints | at 24 weeks
  To evaluate the proportion of eyes with recurrence and the time to recurrence at 24 weeks after the first treatment (recurrence is defined as the recurrence of ridgelike changes or fibrovascular proliferation in the original lesion, complicated by the recurrence of additional lesions in the posterior pole);
Secondary endpoints | within 24 weeks
  To evaluate the proportion of eyes undergoing the second treatment within 24 weeks after the first treatment (the second treatment is defined as the second treatment that is given after the first treatment, regardless of whether the treatment measure is adjusted or not);
Secondary endpoints | within 24 weeks
  To evaluate the proportion of target eyes requiring a second treatment modality within 24 weeks after the first treatment (the treatment modality means laser therapy, anti-VEGF drug therapy and surgery, and the second treatment modality includes change of anti-VEGF drug);
Secondary endpoints | within 24 weeks
  To evaluate the proportion of target eyes whose treatment measures were switched within 24 weeks after the first treatment (the switching treatment is defined as the conversion to laser therapy, anti-VEGF drug therapy and surgery);
Secondary endpoints | within 24 weeks
  To evaluate the number of treatments with Conbercept, ranibizumab, and laser within 24 weeks after the first treatment;
Secondary endpoints | within 24 weeks
  To evaluate the proportion of eyes with ocular AEs within 24 weeks after the first treatment;
Secondary endpoints | within 24 weeks
  To evaluate the proportion of eyes with TEAEs within 24 weeks after the first treatment;
Secondary endpoints | at 24 weeks
  To evaluate the proportion of eyes with aggravated retinopathy staging at 24 weeks after the first treatment;
Secondary endpoints | within 24 weeks
  To evaluate the incidence of endophthalmitis within 24 weeks after the first treatment;
Secondary endpoints | within 24 weeks
  To evaluate the proportion of eyes undergoing vitreous surgery within 24 weeks after the first treatment;
Secondary endpoints | within 24 weeks
  To evaluate the proportion of eyes with ROP complications within 24 weeks after the first treatment. (Complications include cataracts, glaucoma, vitreous hemorrhage, retinal detachment, fibrosis, and ocular atrophy, etc.)

OTHER OUTCOMES:
Exploratory Endpoints | January 1, 2005 to December 31, 2021
  To explore and evaluate the changes in the following longterm observational indicators, which are for descriptive analysis only.
  1、Proportion of target eyes with complete retinal vascularization (the complete retinal vascularization is defined as retinal blood vessels extending to the serrata on the nasal side, and 1 optic disc diameter from the serrata on the temporal side);
Exploratory Endpoints | January 1, 2005 to December 31, 2021
  2. Proportion of eyes with refractive abnormalities;
Exploratory Endpoints | January 1, 2005 to December 31, 2021
  3、Proportion of eyes with abnormal ocular visual function (the ocular visual function indicators include peripheral visual field, etc.);
Exploratory Endpoints | January 1, 2005 to December 31, 2021
  4、Proportion of target eyes with abnormal biological feature (the biological feature include axial length, anterior chamber depth, lens thickness, etc.).

CONTACTS AND LOCATIONS:
Overall Officials: Jianhong Liang, Principal Investigator — Peking University People's Hospital
Locations (2):
- China (2):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: Undecided